CLINICAL TRIAL: NCT02956278
Title: The Effects of BCRP Q141K on Allopurinol Pharmacokinetics and Dynamics
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH); Open Medicine Institute (Unknown)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 14-14550; R01DK103729 (NIH)
Record Dates: First submitted 2016-11-02; First posted 2016-11-07 (Estimated); Results first posted 2020-06-23 (Actual); Last update posted 2020-06-23 (Actual); Status verified 2020-06

CONDITIONS: Chronic Gout; Hyperuricemia
Keywords: allopurinol
MeSH Terms: conditions — Hyperuricemia | interventions — Allopurinol

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- BCRP Q141K CC (Placebo Comparator): Participants that are homozygous reference for BCRP Q141K receive at least one 300 mg dose of allopurinol followed by blood/urine collection for up to 72 hours post-dose.
  Interventions: Drug: Allopurinol; Other: Placebo
- BCRP Q141K CA (Experimental): Participants that are heterozygous for the BCRP Q141K allele receive at least one 300 mg dose of allopurinol, with blood/urine collections up to 72 hours post-dose.
  Interventions: Drug: Allopurinol; Other: Placebo
- BCRP Q141K AA (Experimental): Participants homozygous for the BCRP Q141K allele receive at least one 300 mg dose of allopurinol with blood/urine collection for up to 72 hours post-dose.
  Interventions: Drug: Allopurinol; Other: Placebo

INTERVENTIONS:
Drug: Allopurinol
  Other Names: Zyloprim; Aloprim
Other: Placebo — lactose placebo pill

SUMMARY:
Subjects will undergo a placebo and allopurinol phase to better understand the effects of the reduced function BCRP Q141K variant on allopurinol pharmacokinetics and pharmacodynamics.

ELIGIBILITY:
Inclusion Criteria:

* self-identified as Asian/European ancestry
* generally healthy with approved lab values for CBC,HFP,RFP, and uric acid
* Subjects with the ABCG2 genotype, homozygous, heterozygous or homozygous for the major allele of rs2231142 will be recruited

Exclusion Criteria:

* vascular disease
* renal impairment
* medications/supplements that affect uric acid levels
* pregnant or lactating women
* prior history of allergic reaction to allopurinol or testing positive for HLA-B*5801 allele
* risk of urinary or gastric retention or narrow-angle glaucoma
* impaired hepatic function
* evidence of anemia
* evidence or diagnosis of congestive heart failure
* smokers
* subjects with a mutation other than rs2231142 in the ABCG2 genotype
* subjects taking hormonal contraceptives or other hormonal medications
* evidence of recreational drug use as determined by questionnaire

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 27 (Actual)
Dates: Start 2016-11 (Actual); Primary Completion 2018-03 (Actual); Study Completion 2018-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kathleen Giacomini, PhD, Principal Investigator — University of California, San Francisco
Locations (1):
- Open Medicine Institute, Mountain View, California, United States

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: As the intent of the protocol was to characterize the effect of the genetic variant, data were collected and analyzed per genotype variant regardless of number of doses received.
Groups:
- BCRP Q141K CC: Participants that are homozygous reference for BCRP Q141K receive one 300 mg dose of allopurinol followed by blood/urine collection for up to 72 hours.
- BCRP Q141K CA: Participants that are heterozygous for the BCRP Q141K allele receive one 300 mg dose of allopurinol, with blood/urine collections up to 72 hours.
- BCRP Q141K AA: Participants homozygous for the BCRP Q141K allele receive one 300 mg dose of allopurinol with blood/urine collection for up to 72 hours.
Period: Overall Study
Arm/Group | BCRP Q141K CC | BCRP Q141K CA | BCRP Q141K AA
Started | 15 | 9 | 3
Completed | 9 | 7 | 3
Not Completed | 6 | 2 | 0
Not completed — Withdrawal by Subject | 6 | 2 | 0

BASELINE CHARACTERISTICS:
Population: Subjects were analyzed based on their BCRP Q141K genotype no matter which protocol (single or multiple dose) they participated in.
Groups:
- BCRP Q141K CC Genotype: All subjects that completed the protocol with the reference BCRP Q141K genotype (CC alleles)
- BCRP Q141K CA Genotype: All subjects that completed the protocol with the heterozygous BCRP Q141K genotype (CA alleles)
- BCRP Q141K AA Genotype: All subjects that completed the protocol with the homozygous BCRP Q141K genotype (AA alleles)
- Total: Total of all reporting groups
Arm/Group | BCRP Q141K CC Genotype | BCRP Q141K CA Genotype | BCRP Q141K AA Genotype | Total
Number analyzed (Participants) | 9 | 7 | 3 | 19
Age, Continuous [Mean (Standard Deviation); unit: years] | 26.9 (5.7) | 29.0 (7.2) | 27.3 (6.5) | 27.7 (6.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 1 | 1 | 7
  Male | 4 | 6 | 2 | 12
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 6 | 7 | 2 | 15
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0
  White | 1 | 0 | 0 | 1
  More than one race | 2 | 0 | 1 | 3
  Unknown or Not Reported | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Oxypurinol Renal Clearance
Description: Renal clearance as defined by amount excreted in 24 hours/AUC from 0-24 hours
Time Frame: 24 hours (Urine collected 0-4 hrs,4-8 hrs,8-10 hrs,10-24 hrs post-dose)
Measure: Mean (Standard Deviation); unit: L/hr
Arm/Group | BCRP Q141K CC Genotype | BCRP Q141K CA Genotype | BCRP Q141K AA Genotype
Number analyzed (Participants) | 9 | 7 | 3
L/hr | 1.9 (1.2) | 1.4 (0.5) | 1.6 (0.9)

2. Primary Outcome: Percent Change Uric Acid
Description: Maximum percent change in uric acid after a single dose of allopurinol
Time Frame: 24 hours
Population: Baseline and minimum SUA level after a single dose of allopurinol (i.e. Day 1) were used for the calculation (baseline-minimum)/baseline)
Measure: Mean (Standard Deviation); unit: Percent Change from Baseline
Arm/Group | BCRP Q141K CC Genotype | BCRP Q141K CA Genotype | BCRP Q141K AA Genotype
Number analyzed (Participants) | 9 | 7 | 3
Percent Change from Baseline | 26.8 (5.9) | 23.8 (7.0) | 21.4 (2.5)

3. Secondary Outcome: Oxypurinol AUC
Description: Area under the concentration time curve from 0-24 hours following a single dose of allopurinol (i.e. Day 1 of both protocols)
Time Frame: 24 hours (Collections at 0, 0.5, 1, 1.5, 2, 3, 4, 5, 6, 8, 10, 24 hours post-dose)
Measure: Mean (Standard Deviation); unit: mcg*hr/mL
Arm/Group | BCRP Q141K CC Genotype | BCRP Q141K CA Genotype | BCRP Q141K AA Genotype
Number analyzed (Participants) | 9 | 7 | 3
mcg*hr/mL | 95.9 (25.1) | 99.1 (30.1) | 108.5 (36.1)

ADVERSE EVENTS:
Time Frame: During the course of the protocol and up to 72 hours following the final dose of allopurinol
Groups:
- BCRP Q141K CC: Participants homozygous reference for BCRP Q141K receive one 300 mg dose of allopurinol followed by blood/urine collection for up to 72 hours.
- BCRP Q141K CA: Participants heterozygous for BCRP Q141Kr eceive one 300 mg dose of allopurinol followed by blood/urine collection for up to 72 hours.
- BCRP Q141K AA: Participants homozygous for BCRP Q141Kr eceive one 300 mg dose of allopurinol followed by blood/urine collection for up to 72 hours.
Arm/Group | BCRP Q141K CC | BCRP Q141K CA | BCRP Q141K AA
All-Cause Mortality (participants affected / at risk) | 0/15 | 0/9 | 0/3
Serious Adverse Events (participants affected / at risk) | 0/15 | 0/9 | 0/3
Other Adverse Events (participants affected / at risk) | 0/15 | 0/9 | 0/3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan: Single Dose Protocol (2017-11-07): https://cdn.clinicaltrials.gov/large-docs/78/NCT02956278/Prot_SAP_000.pdf
  • Study Protocol and Statistical Analysis Plan: Multiple Dose Protocol (2017-09-01): https://cdn.clinicaltrials.gov/large-docs/78/NCT02956278/Prot_SAP_001.pdf